CLINICAL TRIAL: NCT07035899
Title: Association of Maternal and Neonatal Umbilical Cord Blood Levels of Propofol Administered for Induction of General Anesthesia With Perinatal Findings in Gravidas Undergoing Cesarean Section
Brief Title: Propofol Anesthesia and Perinatal Outcome
Acronym: PA-Perinatal-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Yilmaz Guler, Obstetric Anesthesia Specialist, Haseki Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PA-PN-O2024
Record Dates: First submitted 2025-05-07; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Complications; Anesthesia
Keywords: Propofol; Pregnancy; Cesarean delivery; Perinatol outcome
MeSH Terms: conditions — Pregnancy Complications | interventions — Cesarean Section

STUDY DESIGN:
Intervention Model Description: Observational
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with Healthy Pregnance undergone Caesarean Section (Sham Comparator): Healthy Pregnant Women between the ages of 18 and 40
  Interventions: Drug: Caesarean Section
- Women Compliceted Pregnance undergone Caesarean Section (Active Comparator): Pregnant women between the ages of 18-40 with Pearclampsia, Preterm Labor, Fetal Growth Retardation, Gestational Diabetes
  Interventions: Drug: Caesarean Section

INTERVENTIONS:
Drug: Caesarean Section — Cesarean section was performed as routine surgical procedure

SUMMARY:
The effects of intravenous propofol administration for general anesthesia in cesarean deliveries on maternal and infant health will be evaluated in relation to maternal and umbilical cord blood propofol levels.

DETAILED DESCRIPTION:
After the ethics committee approval was obtained, volunteers who met the criteria for inclusion in the study were included in the study after obtaining their written permission. After the patients were taken to the operating room, IV catheterization was achieved after CTA, TA and sPO2 monitoring, and the patient was intubated 2 minutes after induction of propfol at 3 mg/kg and rocuronium at 0.6 mg/kg. After the baby was born, an intravenous blood sample was taken from the umbilical cord and the mother simultaneously. After the venous blood samples were obtained as 3 μL, the serum samples obtained by centrifugation as standard were portioned in equal volume to 500 μL Eppendorf tubes and stored at -80°C. After this pre-treatment, propofol was subjected to measurement tests with HPLC, and the collected data were added

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant in ASA category 1-2
* >39 weeks of healthy pregnancy
* >28 weeks complicated pregnancy
* Cesarean delivery with or without action
* Providing induction of general anesthesia with intravenous propofol

Exclusion Criteria:

* Pregnant women under the age of 18,
* Those who have stillbirth,
* Severe chronic kidney and liver disease,
* Neurological disease
* Those with other systemic diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 102 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Blood propofol concentration | The first 5 minutes of cesarean delivery
  ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Sultangazi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No